CLINICAL TRIAL: NCT04492735
Title: The Use of Indocyanine Green as a Diagnostic Adjunct for Pediatric Solid
Brief Title: The Use of Indocyanine Green as a Diagnostic Adjunct for Pediatric Solid Malignancies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Roshni Dasgupta (Other)
Responsible Party: Sponsor-Investigator, Roshni Dasgupta, Roshni Dasgupta, MD, Children's Hospital Medical Center, Cincinnati
Organization: Children's Hospital Medical Center, Cincinnati (Other)
Other Study IDs: PSORC ICG
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Metastatic Disease; Primary Tumor; Solid Malignancies
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Use of indocyanine green will augment the accuracy of identification and resection of both primary solid malignancies as well as their pulmonary metastases, where applicable We will conduct a prospective feasibility study of pediatric patients with solid malignancies with or without lung metastatases who present at the time of initial diagnosis or relapse. These patients will receive a targeted dye to aid in the resection of these metastases. We plan to assess ICG as it relates to:

1. Diagnostic accuracy using pathologic correlation as gold standard measure
2. Short and long term event free and overall survival

DETAILED DESCRIPTION:
Patients diagnosed with solid malignancies or metastatic lesions who require clinically indicated resection will be identified by their Oncologist. The oncologist will inform the subject/family about the study and ask if they may be interested in participating. If the subject/family demonstrates potential interest in the study, the Pediatric Surgery Research team will discuss the risks and benefits of pre-operative ICG administration with the patients and enrollment.

Study subjects: All patients diagnosed with solid malignancies as well as those with metastatic disease distant from the primary tumor will be potentially eligible for the study. Diagnosis will be made:

1. In a multimodal fashion including physical exam, radiologic evaluation (ultrasound, MRI, CT scan, etc), and sometimes biopsy.
2. Prior to definitive surgical resection of the newly diagnosed malignancy

ELIGIBILITY:
Inclusion Criteria:

All patients with newly diagnosed solid, primary malignancies or their related metastatic lesions.

Diagnosis of primary or metastatic malignancy will be made by combination of:

1. Clinical evaluation and physical exam
2. Radiologic study including ultrasound, CT scan, and/or MRI
3. Pathologic diagnosis after biopsy

Exclusion Criteria:

1. Those patients and parents/guardians unwilling to provide consent/assent.
2. Pregnant and/or women who are breast feeding.
3. Patients with Iodine allergies

Ages: 1 Day to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Oncology solid, primary malignancies or their related metastatic lesion
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2020-06-05 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy using pathologic correlation as gold standard measure | 2 years
Short and long term event free and overall survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided